CLINICAL TRIAL: NCT05699070
Title: An Open-label Phase 1 Study to Evaluate Pharmacokinetic/Pharmacodynamic Drug-drug Interactions and Safety/Tolerability of DWC202211 and DWC202212 Compared to Coadministration in Healthy
Brief Title: Drug-drug Interactions Between DWC202211 and DWC202212 in Healthy Subjects
Acronym: DWJ1610
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1610101
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-01

CONDITIONS: Drug-drug Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWC202211 (Experimental)
  Interventions: Drug: DWC202211 100mg
- DWC202212 (Experimental)
  Interventions: Drug: DWC202212 5mg
- DWC202211 + DWC202212 (Experimental)
  Interventions: Drug: DWC202211 100mg + DWC202212 5mg

INTERVENTIONS:
Drug: DWC202211 100mg — DWC202211 for 5 days
  Aspirin 100mg
  Arms: DWC202211
Drug: DWC202212 5mg — DWC202212 for 3 days
  Rabeprazole 5mg
  Arms: DWC202212
Drug: DWC202211 100mg + DWC202212 5mg — DWC202211 + DWC202212 for 5 days
  Aspirin 100mg, Rabeprazole 5mg
  Arms: DWC202211 + DWC202212

SUMMARY:
An open-label phase 1 study to evaluate pharmacokinetic/pharmacodynamic drug-drug interactions and safety/tolerability of DWC202211 and DWC202212 compared to coadministration in healthy

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 50 years at screening
* Subjects with a body weight ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 27.0 kg/m2 at screening

  ※ BMI (kg/m2) = body weight (kg)/[height (m)]2
* Subjects who voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a sufficient explanation on this study and fully understanding the information
* Subjects who are eligible to participate in the study at the discretion of the investigator by physical examination, laboratory tests, and investigator questioning, etc.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04-24 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 27 days
AUClast | up to 27 days

SECONDARY OUTCOMES:
DWC202211 Tmax,ss | up to 27 days
DWC202211 T1/2,ss | up to 27 days
DWC202211 Cmin,ss | up to 27 days
DWC202211 Cavg,ss | up to 27 days
DWC202211 CLss/F | up to 27 days
DWC202211 Vdss/f | up to 27 days
DWC202211 PTF | up to 27 days
DWC202212 Tmax,ss | up to 27 days
DWC202212 T1/2,ss | up to 27 days
DWC202212 Cmin,ss | up to 27 days
DWC202212 Cavg,ss | up to 27 days
DWC202212 CLss/F | up to 27 days
DWC202212 Vdss/f | up to 27 days
DWC202212 PTF | up to 27 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea